CLINICAL TRIAL: NCT04680871
Title: Validation of In-Ear Sensor
Status: Withdrawn | Type: Observational
Why Stopped: Study not being pursued
Sponsor: Starkey Laboratories, Inc (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PR 2020-409
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2020-12

CONDITIONS: Biometrics Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Normal, Healthy Subjects
  Interventions: Device: In-Ear Sensor
- Induced Febrile Subjects
  Interventions: Device: In-Ear Sensor

INTERVENTIONS:
Device: In-Ear Sensor — The device will passively monitor participants' biometrics

SUMMARY:
The purpose of this study is to clinically validate noninvasive in-ear sensor.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is an adult over 18 years of age (18 to 50 for Induced Febrile Subjects)
* Subject must be willing and able to comply with study procedures and duration. Subject must be willing and able to comply with study procedures and duration. Must be available for at least 2 visits for ear molds and study conduct.
* Male or female of any race

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant or who have a urine test positive for pregnancy on the day of the study (For Induced Febrile Subjects only)
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * Resting high blood pressure: systolic >140 mmHg or diastolic >90 mmHg on 3 consecutive readings (For Induced Febrile Subjects only)
  * have had cardiovascular surgery
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * thyroid disease (controlled and uncontrolled)
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * Cancer / chemotherapy
* Subjects with medical inflammatory conditions/taking antiinflammation medications

  * Barbiturates
  * Antipsychotics
  * Recent immunizations (within 1 month)
  * Subjects who have taken antipyretics in the last 240 minutes (aspirin, acetaminophen, ibuprofen)
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will involve healthy participants 18-50 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Biometric | 1-2 months
  Biometric data collected from in-ear sensor device and compared to validated reference device

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No